CLINICAL TRIAL: NCT04536883
Title: Contribution of Confocal Microscopy in the Diagnosis of Acute Cell Rejection ACR in Lung Transplantation: Pilot Study
Brief Title: MICRA - Pilot Study
Acronym: MICRA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nantes University Hospital (Other)
Collaborators: Institut de Recherche en Santé Respiratoire des Pays de la Loire (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: RC20_0201
Record Dates: First submitted 2020-08-24; First posted 2020-09-03 (Actual); Last update posted 2021-10-06 (Actual); Status verified 2021-03

CONDITIONS: Rejection Lung Transplant
Keywords: Confocal Microscopy; Acute cell rejection; Lung Transplantation
MeSH Terms: interventions — Microscopy, Confocal

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Microscopy confocal (Experimental): The fibroscopy is carried out according to the usual procedure of the service. During the fibroscopy, for all patient, the confocal microscopy procedure begins.
  After the end of confocal procedure, 5 to 6 transbronchial biopsies are performing
  Interventions: Procedure: microscopy confocal

INTERVENTIONS:
Procedure: microscopy confocal — At this stage, the confocal microscopy procedure begins:
  Taking pictures for post-procedure analysis in 4 different territories. For each territory, the investigator need to get a snapshot of a vascular structure and a snapshot of an alveolus.
  Analysis per procedure: the same operator analyzes the alveoli deemed to be representative in real time. It determines the presence of intra-alveolar inflammatory cells and answers the question of the main criterion: possible interpretation in confocal microscopy? YES / NO, the clinical researcher immediately notes the answer in the CRF. Based on this per-procedure analysis, if he deems the interpretation possible, the operator declares if he concludes that pulmonary inflammation is present YES / NO, the response is noted immediately in the CRF.
  The fibroscopy procedure is then resumed as usual in the department, namely:

SUMMARY:
Acute cell rejection is a common complication of lung transplantation. The pathological diagnosis is based on the performance of transbronchial biopsies which are associated with a significant risk of potentially severe pneumothorax and hemoptysis. Confocal microscopy performed during bronchial endoscopy provides real-time images of the lungs on a microscopic scale. Thus, it is possible to visualize the alveoli, capillaries and intra-alveolar inflammatory cells. So far, work on the subject has only investigated the ability of this technique to determine the presence of acute cell rejection on post-fibroscopy analysis. Our hypothesis is that the absence of airway inflammation seen during the procedure by confocal microscopy is able to rule out the diagnosis of ACR and avoid the performance of transbronchial biopsies. Our job is to first assess the feasibility of the per-procedure evaluation and determine a decision algorithm. If the result is conclusive, a larger study will be carried out to assess the negative predictive value of this approach for the diagnosis of acute cell rejection.

DETAILED DESCRIPTION:
During the patient's usual follow-up, if an ACR is suspected and it is decided to perform an endoscopy with transbronchial biopsies, the protocol is presented to the patient by the doctor in charge. If the patient agrees to participate in the study, consent is obtained. Collection on arrival of the patient's sex, age, weight, height, respiratory background leading to the patient's lung transplant.

According to the department's protocol: carrying out functional respiratory tests, a biological assessment (CBC, hemostasis and CRP) and a chest x-ray prior to the procedure except if there is another chest imaging dating less than 24 hours testifying to the absence of pneumothorax. Premedication with hydroxyzine, insertion of a peripheral venous route, verification of the patient's identity, anticoagulant or anti-aggregating treatment and potential allergy.

The fibroscopy is carried out according to the usual procedure of the service, namely: realization of 1 to 2 mg of hypnovel intravenously depending on the patient's tolerance, introduction of the fiberscope preferably via the nasal route, if impossible or contraindicated, the oral route is possible with the use of a bite block to protect the fiberscope. Visualization of the mobility of the vocal cords, trachea, carina and right and left bronchial tree up to the segmental level. Identification of the quality of the sutures and the possible presence of bronchial stenosis. Realization of a bronchial trap with bacteriological and mycological analysis. Performing a bronchoalveolar lavage (90cc of physiological serum, preferably in the middle lobe) with anatomopathological, virological, bacteriological, mycological and mycobacteriological analysis.

At this stage, the confocal microscopy procedure begins:

Taking pictures for post-procedure analysis in 4 different territories. For each territory, the investigator need to get a snapshot of a vascular structure and a snapshot of an alveolus.

Analysis per procedure: the same operator analyzes the alveoli deemed to be representative in real time. It determines the presence of intra-alveolar inflammatory cells and answers the question of the main criterion: possible interpretation in confocal microscopy? YES / NO, the clinical researcher immediately notes the answer in the CRF. Based on this per-procedure analysis, if he deems the interpretation possible, the operator declares if he concludes that pulmonary inflammation is present YES / NO, the response is noted immediately in the CRF.

The fibroscopy procedure is then resumed as usual in the department, namely:

Performing 5 to 6 transbronchial biopsies. The number of biopsies depends on the patient's tolerance and the occurrence of complications such as hemorrhage or pneumothorax. Checking at the end of the procedure for the absence of active intra-bronchial bleeding, followed by a frontal chest X-ray to check for the absence of pneumothorax (examination carried out routinely even in the event of bronchial endoscopy with simple BTB). If there are no complications and if the pathological analysis of the lung biopsies does not conclude that there is an acute cellular rejection, the patient can return home at the end of the day. If the pathologist concludes that there is a rejection or that there is a complication, the patient remains hospitalized for the time necessary for medical treatment.

ELIGIBILITY:
Inclusion Criteria:

* Follow-up by the Nantes University Hospital team for a lung transplant
* Having given their consent
* Clinical suspicion of acute cellular rejection OR systematic fibroscopy post transplantation to screen for acute asymptomatic rejection

Exclusion Criteria:

* Minor or adult patient under guardianship and protected person
* FEV1 <40% of theoretical at the time of inclusion
* Bleeding disorder
* Pneumothorax existing before the performance of the fibroscopy
* Active smoking less than 1 year old

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2020-09-23 (Actual); Primary Completion 2021-08-18 (Actual); Study Completion 2021-08-18 (Actual)

PRIMARY OUTCOMES:
Determine ability of the operator | 1 day
  The main objective of this study is to determine the ability of the operator to obtain and interpret confocal microscopy images per procedure. analyzes in real time the images provided by the confocal microscopy probe. the operator determines the presence of intra-alveolar inflammatory cells and evaluates the vessel wall.
  On the basis of this per-procedure analysis, if the operator considers the interpretation possible, he declares whether he concludes that the presence of pulmonary inflammation is consistent with the diagnosis of rejection.

SECONDARY OUTCOMES:
Adverse effects | 1 day
  assess the adverse effects: patient comfort, procedure time and complications (hemoptysis, pneumothorax
ability of confocal microscopy to eliminate acute cellular rejection | 1 day
  assess the ability of confocal microscopy to eliminate acute cellular rejection
Correlation confocal microscopy and proven infection | 1 day
  to assess the correlation of the parameters observed in confocal microscopy associated with a proven infection (main differential diagnosis of acute cell rejection)
Correlation inter operator | 1 day
  The correlation between the analysis per procedure by the operator and the analysis of the images by the second a posteriori expert

CONTACTS AND LOCATIONS:
Overall Officials: Adrien TISSOT, MD, Principal Investigator — Nantes University Hospital
Locations (1):
- CHU Nantes, Nantes, France

IPD SHARING:
Plan to Share IPD: Undecided